CLINICAL TRIAL: NCT02059538
Title: Metagenomics and Integrative Systems Medicine of Cardiometabolic Diseases
Acronym: METACARDIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P121102; IDRCB2013-A00189-36 (Other: IDRCB Number)
Record Dates: First submitted 2013-11-07; First posted 2014-02-11 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2013-06

CONDITIONS: Cardiometabolic Disease
Keywords: Obesity; Type 2 diabetes; Coronary artery diseases; Microbiota; Omics (ie transcriptomics, metabolomics, metagenomics, lipidomics)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Injections, Subcutaneous; Liver Extracts; Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1 (Other): Metabolic syndrome
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 2 (Other): Severly obese patients
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 3 (Other): Type-2 diabetics patients
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 4 (Other): Patients with first recent (< 2 weeks) acute coronary syndrome (ACS)
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 5 (Other): Patients with stable chronic coronary artery disease without heart failure
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 6 (Other): Patients with ischemic systolic heart failure (CHF)
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 7 (Other): Patients with non-ischemic chronic heart failure
  Interventions: Other: Adipose tissue biopsies (omental and subcutaneous) liver; Radiation: CT-scan; Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)
- Group 8 (Other): Healthy volunteers
  Interventions: Other: Stools sampling; Other: DNA sampling; Other: Blood sampling; Other: Urine sampling; Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)

INTERVENTIONS:
Other: Adipose tissue biopsies (omental and subcutaneous) liver
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7
Radiation: CT-scan
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7
Other: Stools sampling
Other: DNA sampling
Other: Blood sampling
Other: Urine sampling
Radiation: Dual energy X-ray absorptiometry-scan (DEXA-scan)

SUMMARY:
Supported by state-of-the-art systems medicine competences including integrative computational and functional genomics, the overarching goal of the trial is to investigate the impact of qualitative and quantitative changes in the gut microbiota on the pathogenesis of cardiometabolic diseases (CMDs) and their associated co-morbidities. A major objective will be to translate the clinical and fundamental based discoveries into new diagnosis and preventive actions paving the way to novel modes of treatment in the successive stages of CMD progression.

DETAILED DESCRIPTION:
Cardiovascular diseases represent a huge medico-economic issue that is supported by public health policy. It is linked not only to the high prevalence of these diseases but also the associated cost they encounter for. Therefore, it seems rather urgent to create and validate tools to predict evolution of this group of disease in order to better take care of patients before they enter the more chronic stages which induce increased costs and socioeconomic and medical burdens.

It is now well acknowledged that gut microbiota is modified in some metabolic disease such as type-2 diabetes but also in inflammatory diseases. However, gut microbiota is still insufficiently explored in cardiovascular disease, although it could represent a useful, non-invasive and practical tool in the daily care of patients.

Investigators aim to deepen the knowledge and characterization of gut microbiota in patients going from metabolic diseases such as metabolic syndrome, obesity and type 2 diabetes (which are risks factors for cardiovascular diseases) to overt coronary artery diseases (from the first event to end stage heart failure). Investigators will use a system medicine approach whose aim is to integrate numerous data coming from different technologies (including environment, transcriptomics, metabolomics, metagenomics, lipidomics and bioinformatics). These integrated approaches are needed to translate basic science findings into clinical practice for the benefit of the patients.

Investigators aim to uncover new microbial signatures that could help diagnose and/or predict both the natural evolution of cardiometabolic diseases and the response to treatment. Investigators aim to go forward personalized medicine.

Patients will be approached for enrolment during their hospitalization in the 3 centers during the 24-month enrolment phase (WP3). Once the informed consent completed, each patient will be assessed for CMD phenotypes including clinical examination, environmental and food habit evaluation, blood urine and feces samples. In each group of patients, a sub-sample of 30 to 50 subjects will be included in one or more advanced phenotyping items. This will include whole body composition by absorptiometry (DXA), abdominal visceral fat by tomodensitometry, Oral Glucose Tolerance Test (OGTT) (glucose, insulin, incretins), subcutaneous fat biopsy, cardiac echocardiography, intima media thickness, pulse wave velocity. For the obese patients undergoing bariatric surgery: liver and subcutaneous and omental adipose tissue biopsies will be obtained during surgery.

This group of patient will be followed at 3, 6 and 12 months after their surgery and will have the same examination as mentioned above.

ELIGIBILITY:
Inclusion criteria :

Group 1 : metabolic syndrome As defined by the IDF

* Central obesity: defined as waist circumference > 94 cm for European men and > 80 cm for European women (with knowledge on ethnicity for other groups)
* plus 2 of the following criteria out of 4:

  * Elevated blood pressure with systolic ≥ 130 mmHg and/or diastolic ≥85 mmHg (or patients receiving anti-hypertensive drug treatment)
  * Triglycerides ≥1.50mg/dl (1.71mmol/l) (or patients receiving drug treatment for elevated triglycerides)
  * HDL-c<40mg/dl (1.03 mmol/l) in males or HDL-c<50mg/dl (1.29mmol/l) in females (or patients receiving drug treatment that reduces HDL-c)
  * Elevated fasting glucose: Glycemia ≥100mg/dl
* Aged 18 to 75 years old

To avoid overlapping with the other groups (in particular group III): only patients with normal glucose tolerance (NGT), impaired glucose tolerance (IGT) and/or impaired fasting glucose (IFG) and an HbA1c < 6.5 % will be included in this group.

Group II: severely Obese patients

* Aged 18 to 75 years old
* BMI ≥35kg/m²
* Half of the effective will be standard obese patients (150 in Paris and 150 in Leipzig)
* Half of the effective will be patients candidate to a bariatric surgery either Sleeve gastrectomy or Roux-en-Y bypass (with the following clinical conditions: according to European and national guidelines for obesity surgery):

  * BMI ≥40 kg/m² or
  * BMI ≥35kg/m² with at least 1 obesity-related comorbidity (Hypertension, dyslipidemia, obstructive sleep apnea, joints disease and even type 2 diabetes).those can have past history of coronary diseases.

These patients will be followed during the first year after surgery. The clinical and research investigation time points will be 3, 6 and 12 months after the surgery.

Group 3: type 2 diabetes

Patients with known type 2 diabetes ie:

* Fasting plasma glucose (FPG) ≥7 mM (=1.26g/l) without treatment or Patients with HbA1c ≥ 6.5% (48 mmol/mol) without treatment or Patients treated with any anti diabetic agent whatever the HbA1c level at the day of the study <10%
* BMI ≥ 25kg/m²
* No symptomatic CAD and previous CVD events
* with all stages of albuminuria
* Aged 18-75 years old

Group 4

- Aged 18-75 years ACS without persistent ST elevation (ST-) Or ACS with persistent ST elevation (STEMI)

Group 5

* Aged 18-75 years
* Stable CAD is defined by
* CAD:ie (Previous documented ACS or previous coronary dilatation >6 months or previous planned PCI showing a significant CAD (coronary stenosis > 30 % in at least on major coronary artery) leading or not to a PCI / stent implantation) and Stable ie: (previous surgical coronary revascularization (CABG > 6 month) or no symptoms or stable angina for 6 months and Without heart failure ie: (Left ventricular ejection fraction ≥ 45 %)

Group 6 Part of this group will be recruited during or immediately after a hospitalization for acute heart failure and Another part of the group will be at the stage in chronic heart failure with no recent acute event (no acute decompensation < 3 month)

chronic Cardiac disease :ie Duration of chronic heart failure > 6 months, or NYHA 2-4 or past history of clinical insufficiency decompensation or CHF due to LV systolic dysfunction (LV ejection fraction < 45 %) and Past history of ACS and /or documented CAD ie (stenosis > 30 % in > 1 coronary artery or previous revascularization >6months) and Aged 18 to 75 years old

Group 7 Half of this group will be recruited during or immediately after a hospitalization for acute heart failure (< 1 month) and half in chronic stable heart failure (no acute decompensation < 3 month) chronic cardiac disease non ischemic ie: (Documented coronary angiogram showing non-significant CAD) cardiac insufficiency ie: (LV ejection fraction < 45 %, or NYHA 2-4 or past history of clinical insufficiency decompensation) and No valvular etiology and No symptoms and no angina and Aged 18 to 75 years old Group 8

* Age and sex matched to the patients cohorts
* Lean (19kg/m² < BMI <25 kg/m²)
* Aged 18 to 75 years old

Exclusion criteria :

Definitive exclusion criteria:

* <18 or >75 years old
* Past history of abdominal cancer+/- radiation therapy on the abdomen
* past history of intestinal resection except for appendicectomy
* Participants with acute or chronic inflammatory or infectious diseases (including VHC, VHB and HIV)
* Organ transplantation
* Patient on Immunosuppressive therapy
* Patients with severe kidney failure and or patients on dialysis therapy or eGFR < 50 ml/min per 1.73 m2 body surface area)
* Non affiliated to social security
* Patients who do not understand the research procedures or those that are institutionalized, or those unable to give informed consent
* Patients who decline participation
* Patients with drug or alcohol addiction

Temporary exclusion criteria:

* Recent lost of weight >10 kilos in the past 3 months
* Recent antibiotic treatment (<2months)
* Patients on non-steroid anti-inflammatory treatment for the past 48 hours
* Patients on laxative therapy that could modify the bowel transit in the past week
* Patients on therapy that can modify transit time (orlistat and acarbose)
* Pregnant women or breast feeding women
* Patients who are already included in a clinical study which implies testing any pharmaceutical drug. On the other hand, patients recruited in other observational studies can be recruited in METACARDIS

Specific exclusion criteria per group Group I : Type-2 diabetic patients or patients on anti-diabetic agent Clinical signs of CAD Past history of coronary syndrome

Group II : Obese

IIa:

Type 2 diabetic patients Past history of coronary syndrome Clinical signs of CAD

IIb:

Patients with previous bariatric surgery

Group III Past history of coronary syndrome Clinical signs of CAD Known auto-immune diabetes mellitus Patients with a HbA1c > 10 % We will exclude secondary diabetes mellitus or type 1 or Idiopathic diabetes or Other specific types of diabetes Genetic defects of the β-cell or Genetic defects in insulin action or Diseases of the exocrine pancreas or Endocrinopathies or Drug- or chemical-induced diabetes or diabetes due to pancreatic resection

Group IV Past history of coronary syndrome Left ventricular dysfunction FeVG<45%

Group V Left ventricular dysfunction FeVG<45%

Group VII Significant documented CAD Past history of coronary syndrome

Group VIII Patients with known chronic inflammatory diseases Patients with either type 2 diabetes, cardiovascular diseases, Patients with treatment for dyslipidemia or for hypertension Patients with chronic inflammatory diseases, Patients with diseases of the gastrointestinal tract, including prior major abdominal surgery on the gastrointestinal tract Patients on non-steroid anti-inflammatory treatment or after a wash-up period of 2 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2350 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Look for differences in gut microbiota signatures using metagenomic approach in the 8 different groups | baseline
  Look for differences in gut microbiota signatures using metagenomic approach in the 8 different groups (metabolic syndrome, type 2 diabetes, obesity, acute coronary event, chronic coronaropathy with or without cardiac insufficiency, cardiac insufficiency without coronaropathy and controls), in order to uncover gut derived signature associated with CMD stages

SECONDARY OUTCOMES:
Establish differences in fecal metabolomic signatures using 1H nuclear magnetic resonance (NMR) spectroscopy and Ultra-high Performance Liquid Chromatography Mass Spectrometry ((UPLC-MS) on fecal samples) in the 8 different groups (cf above mentioned) | baseline

OTHER OUTCOMES:
Establish differences in systemic and adipose tissue inflammatory patterns (using multiplex array and adipose tissue transcriptomic) in the 8 above mentioned groups | Baseline
Establish host metabolomic differences in the 8 groups in order to obtain a CMD metabolomic derived signature (using 1H nuclear magnetic resonance) spectroscopy and Ultra-high Performance Liquid Chromatography Mass Spectrometry (in serum and urine) | Baseline
Establish a statistical association between host metabolomic signatures (cf above 3 in serum and urine) and the gut metagenomic signatures in the 8 groups | Baseline
Establish a diet related signature of CMD stages by looking for differences in diet in the 8 groups (using Food Frequency Questionnaire (FFQ) and three day 24h diet recall) | Baseline
Establish an environment related signature of CMD stages by looking at differences in environment in the 8 groups (using data obtained from environment questionnaires) | Baseline
Look for statistical association between gut derived signatures and lifestyle factors such as environment and diet (using data obtained from environment questionnaires and the results of both FFQ and Three day 24h diet recall) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Karine Clement, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- University of Copenhagen, Copenhagen, Denmark
- Hôpital Pitié-Salpétrière, Paris, France
- University of Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Belda E, Voland L, Tremaroli V, Falony G, Adriouch S, Assmann KE, Prifti E, Aron-Wisnewsky J, Debedat J, Le Roy T, Nielsen T, Amouyal C, Andre S, Andreelli F, Bluher M, Chakaroun R, Chilloux J, Coelho LP, Dao MC, Das P, Fellahi S, Forslund S, Galleron N, Hansen TH, Holmes B, Ji B, Krogh Pedersen H, Le P, Le Chatelier E, Lewinter C, Manneras-Holm L, Marquet F, Myridakis A, Pelloux V, Pons N, Quinquis B, Rouault C, Roume H, Salem JE, Sokolovska N, Sondertoft NB, Touch S, Vieira-Silva S; MetaCardis Consortium; Galan P, Holst J, Gotze JP, Kober L, Vestergaard H, Hansen T, Hercberg S, Oppert JM, Nielsen J, Letunic I, Dumas ME, Stumvoll M, Pedersen OB, Bork P, Ehrlich SD, Zucker JD, Backhed F, Raes J, Clement K. Impairment of gut microbial biotin metabolism and host biotin status in severe obesity: effect of biotin and prebiotic supplementation on improved metabolism. Gut. 2022 Dec;71(12):2463-2480. doi: 10.1136/gutjnl-2021-325753. Epub 2022 Jan 11. PMID 35017197